CLINICAL TRIAL: NCT03993743
Title: An Open-label, Dose Escalation Clinical Study to Access the Safety and Clinical Activity of CD147-targeted CART by Hepatic Artery Infusions for Very Advanced Hepatocellular Carcinoma
Brief Title: A Study of CD147-targeted CAR-T by Hepatic Artery Infusions for Very Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chen Zhinan, Director of National Translational Science Center for Molecular Medicine, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chen Zhinan-1
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: liver cancer; CD147; CAR-T
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD147-CART (Experimental): Infusions of CD147-CART cells over the course of each week for 3 times into the hepatic artery
  Interventions: Biological: CD147-CART

INTERVENTIONS:
Biological: CD147-CART — Three infusions of CD147-CART cells over the course of three weeks into the hepatic artery.
  Other Names: anti-CD147 chimeric antigen receptor T cell

SUMMARY:
This is a single-center, single-arm, open label and dose escalation clinical study of anti-CD147 CART cells by hepatic artery infusions in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Patients autologous T cells are activated and then engineered to express chimeric antigen receptors (CARs) specific for CD147(CD147-CART). CAR-T cells are expanded in culture and returned to the patient by hepatic artery infusion at specific cell doses. Four CD147-CART doses patient are planned at 1-week intervals. Tumor biopsies will be obtained at the time of the initial diagnostic angiogram and during the first infusion session. Serum cytokine level and CAR-T cell number will be measured in whole treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 year and ≤ 65 years, both male and female.
2. Advanced hepatocellular carcinoma(HCC) patient, which is untreatable by surgery or local therapy, or has postoperative progressions, failed at least one and two line of standard systemic chemotherapy, and unwilling or intolerance to targeting therapy or immune-therapy of cancer.
3. The portal vein is not total occlusion, or collateral circulation has formed between hepatic artery and blocked portal vein.
4. Patient with measurable HCC focus defined by mRECIST.
5. Patient with histologically confirmed diagnosis of CD147+ hepatocellular carcinoma.
6. Adequate venous access for apheresis, and no other contraindications for apheresis.
7. Child-Pugh score ≤7.
8. Eastern Cooperative Oncology Group(ECOG) performance status of 0-2.
9. Patient with a life expectancy of greater than three months.
10. Patients must able to understand and be willing to sign an informed consent.

Exclusion Criteria:

1. Patients with fibrolamellar carcinoma of liver，mixed hepatocellular carcinoma or cholangiocarcinoma.
2. Patients with severe hypohepatia including jaundice, hepatic encephalopathy, refractory ascites or hepatorenal syndrome.
3. Patients with severe comorbidity, including any of the following.

   1. Unstable angina pectoris and/or congestive heart failure need hospitalization;
   2. Myocardial infarction or cerebrovascular accident (CVA) in the last 6 months;
   3. chronic obstructive pulmonary disease progressions or need hospitalization;
   4. severe cardiovascular, nervous system, hematological, gastrointestinal, endocrine diseases or metabolic disorders;
   5. autoimmune disease or immunodeficiency disease;
   6. acute bacterial infections or fungal infections needs intravenous injection of antibiotics during CAR-T cell therapy;
   7. tuberculosis not cured;
   8. other malignancies;
4. Patients who have received gene therapy, cell therapy or immune therapy.
5. Patients who have received organ transplantation.
6. Patients who have received treatment of targeted drugs, glucocorticoid or immunosuppressive drugs within 2 weeks before enrolling in clinical trial.
7. Patients who have received chemotherapy except for lymphocyte clearance within 2 weeks before enrolling in clinical trial.
8. Patients who have received radiotherapy.
9. Patients who did not recover to CTCAE(v5.0) grade 1 from adverse events （except hair）of previous anti-tumor therapy before enrolling in trial.
10. Syphilis test (TRUST) positive, Anti-HIV positive, Anti-HCV positive with HCV-RNA level higher than the lower limit of detection(LOD), or HBcAb positive with HBV-DNA level higher than the LOD.
11. Patients with following abnormalities:

    1. Absolute neutrophil count (ANC) < 1.5E9/L, platelet(PLT) < 50E9/L, or hemoglobin(HGB)< 80 g/dL;
    2. Prothrombin time (PT), activated partial thromboplastin time (APTT) or international normalized ratio (INR) > 1.5×ULN (upper normal value);
    3. Total bilirubin(TBIL) > 2×ULN; ALT, AST or ALP>5×ULN;
    4. Serum creatinine (Cr)≥1.5×ULN or glomerular filtration rate (GFR) < 60 mL/min·1.73m^2;
    5. left ventricular ejection fraction (LVEF) < 50%;
12. Patients with a history of allergic reactions attributed to any agents or compounds involved in this study.
13. Patients with a history of mental disorders.
14. Patients with a history of drug abuse.
15. Pregnant and lactating women.
16. Patients of childbearing age who unwilling or unable to take birth control from during this study and 3 months post this study.
17. Patients who receive any other investigational agents within the 3 months before enrolling in this clinical trial.
18. Investigator considers not suitable for this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-10-27 (Estimated); Study Completion 2022-05-27 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of adverse events induced by CD147-CART hepatic artery infusions | 12 weeks
  To assess the safety of CD147-CART (anti-CD147 CAR-T cell) hepatic artery infusions (HAI) for very advanced hepatocellular carcinoma which measured by number and type of adverse events.

SECONDARY OUTCOMES:
DLT and MTD of CD147-CART cell hepatic artery infusions | 12 weeks
  To determine the dose limited toxicity (DLT) and maximum tolerated dose (MTD) of CD147-CART hepatic artery infusions.
Activity of CD147-CART cell hepatic artery infusions | 2 years
  To evaluate treatment response of CD147-CART hepatic artery infusions for very advanced hepatocellular carcinoma.
CD147-CART detection in extrahepatic sites | 2 years
  Quantification of CD147-CART cells in blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of hepato-biliary & Pancreato Splenic Surgery Organ Transplant Center, Xijing Hospital, Xi'an, Shaanxi, China